CLINICAL TRIAL: NCT03798964
Title: The Expression Heparanase in Term and Preterm Placentas
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0119-18
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Elective term cesarean: Low-risk women undergoing elective term cesarean section
  Interventions: Other: Placental analysis
- Term vaginal delivery: Low-risk women undergoing term vaginal delivery
  Interventions: Other: Placental analysis
- Preterm vaginal delivery: Women undergoing preterm vaginal delivery
  Interventions: Other: Placental analysis

INTERVENTIONS:
Other: Placental analysis — Analysis of placenta to determine expression of heparanase

SUMMARY:
Heparanase is an endo-β-glucuronidase that cleaves heparin-sulfate (HS) side chains of heparan sulfate proteoglycans, an integral constituent of the extra cellular matrix (ECM).

This study aims to investigate the association between heparanase expression in the human placenta and preterm birth (PTB) .

The investigators hypothesize that an abnormal placentation causes relative placental ischemia that induces higher rates of heparanase expression.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy

Exclusion Criteria:

* High-risk patients
* Multiple pregnancy
* Significant maternal illness
* Significant fetal anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women attending our obstetrical unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Heparanase expression | Six months
  Heparanase expression in the human placenta following delivery will be evaluated by western blot analysis in the three groups and will be compared to determine differences in the levels.

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No